CLINICAL TRIAL: NCT05275361
Title: Pilot Study Utilizing Social Contacts to Facilitate Mammogram Screening Among African American Women
Brief Title: Utilizing Social Contacts to Facilitate Mammogram Screening Among African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202110124
Record Dates: First submitted 2022-02-04; First posted 2022-03-11 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Mammogram; Breast Cancer Screening; African American women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient: Scheduled for mammogram (Experimental): * Will be asked to choose 2 social contacts (adult family member or friend identified by the participant as someone who could be engaged by the research team to encourage the participant to attend her mammogram appointment)
  * Will receive reminder(s) from social contact about the screening mammogram appointment
  * Will receive reminder from Breast Health Center about screening mammogram appointment
  * Will be contacted to provide experience with the study
  Interventions: Behavioral: Social Contact Reminder
- Social Contact of Patient (No Intervention): * Facilitate enrolled patient to complete the screening mammogram.
  * Will receive information about screening mammograms and resources available at the Breast Imaging Center.
  * Will be contacted approximately 3 days prior to the patient's mammogram appointment.
  * Will be contacted to provide experience with the study

INTERVENTIONS:
Behavioral: Social Contact Reminder — -The social contact will remind patient about screening mammogram appointment
  Arms: Patient: Scheduled for mammogram

SUMMARY:
Eliminating racial disparities in breast cancer is a top public health priority. African American (AA) women often present with more advanced and aggressive disease at the time of diagnosis and are more likely to die from breast cancer than any other racial/ethnic group in the United States. Mammogram screening significantly reduces breast cancer mortality by diagnosing cancer at an earlier stage where treatments are more effective. While some AA women do not schedule screening mammograms as recommended by current guidelines, others do not show up for their exams after scheduling them (no-shows). No-shows to cancer screening appointments impose an enormous strain on our limited healthcare resources with negative impact on other patients who could have secured earlier appointments, loss of revenue for hospitals or clinics serving underserved populations and delays in diagnoses and treatment for those who do not have screening. The investigators identified a high no-show rate for screening mammograms at our hospital. AA women were almost three times more likely to no-show for their mammograms compared to White women. Patient's social networks plan an important role in health promotion. In this study, we will pilot an intervention involving patient's social contacts (family, friends, neighbors, etc.) as healthcare facilitators to improve appointment attendance. The investigators seek to determine whether this intervention is feasible and acceptable to patients and whether this intervention will improve attendance rates for screening mammograms among AA women at our institution. If effective, the use of a patient's social contact person as a healthcare facilitator (similar to a patient navigator) would be a readily available and inexpensive resource for other institutions to implement.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Female
* African American
* At least 40 years old
* Scheduled for a screening mammogram within 3 months following initiation of the study
* Willing and able to provide contact information for two adult social contacts (friends or family members)

Exclusion Criteria for Patients:

-Prior history of breast cancer

Inclusion Criteria for Social Contacts:

* At least 18 years old
* Selected by the patient as someone (family member or friend) who would be able to support her in keeping her mammogram appointment

Exclusion Criteria for Social Contacts:

-Less than 18 years of age

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting patients' social contacts to serve as healthcare facilitators as measured by number of participants enrolled to the study with a social contact that agrees to participate | Through completion of enrollment (estimated to be 3 months)
  -The study is deemed feasible if 80 participants are enrolled to the study and further, if at least 65% of the 80 participants will have a social contact agreeing to participate

SECONDARY OUTCOMES:
Describe demographic characteristics of the social contacts and any associations with patient appointment attendance | Through mammogram appointment (estimated to be 6 months)
  -Use descriptive statistics to present the characteristics of social contacts and regression analysis to determine in association with social contact characteristics and appointment attendance.
Rate of mammography attendance | Through mammogram appointment (estimated to be 6 months)
Using a structured survey interview, determine the percentage of patients and their social contacts who respond positively (agree or strongly agree) that the intervention helped them keep their scheduled screening mammogram appointment | Through mammogram appointment (estimated to be 6 months)
  -Use descriptive statistics to present response to structured interview questions.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Hensing, M.D., M.S., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu